CLINICAL TRIAL: NCT00062439
Title: A Phase II Trial of Induction Chemoradiotherapy With Cisplatin/Etoposide Followed by Surgical Resection, Followed by Docetaxel, for Non-Small Cell Lung Cancer Involving the Superior Sulcus (Pancoast Tumors)
Brief Title: S0220: Chemoradiotherapy Followed By Surgery and Docetaxel in Treating Patients With Pancoast Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); American College of Surgeons (Other); North Central Cancer Treatment Group (Network); NCIC Clinical Trials Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304777; U10CA032102 (NIH); S0220 (Other: SWOG)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etoposide, Cisplatin, Thoracic RT, Surgery, Docetaxel (Experimental)
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: etoposide; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — During induction:50 mg/m2,IV on Days 1, 8, 29 & 36. In any appropriate vehicle over 60 minutes
Drug: docetaxel — During consolidation: 75 mg/m2 IV on Day 1, every 21 days for 3 cycles over 60 minutes
Drug: etoposide — During induction: 50 mg/m2, IV on Days 1 - 5 Days 29 - 33. In 250 ml of NS over 60 minutes.
Procedure: conventional surgery — If, based upon the evaluation in Section 7.4a, there is no evidence of progression (see Section 10.2d for definition), patients will proceed to the next appropriate step: Registration #2 and surgery followed by Registration #3 and additional chemotherapy (Sections 7.5 and 7.6). Response determinations (CR,PR, SD) will be required. If criteria for progressive measurable or nonmeasurable disease (see Section 10.0) are met, the patient will then be removed from protocol treatment and receive follow-up according to the schedule. Surgery will be performed 3 - 7 weeks after completion of chemoradiotherapy.
Radiation: radiation therapy — Radiotherapy is to begin within 24 hours following the start of chemotherapy. Day 1 of radiotherapy must be a Monday, Tuesday or Wednesday, but no later in the week to insure simultaneous therapy for the majority of each chemotherapy cycle. The total dose to the prescription point will be 4,500 cGy given in 25 fractions. The patient will be treated with one fraction per day with all fields treated per day. 180 cGy will be delivered to the isocenter.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, etoposide, and docetaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining cisplatin and etoposide with radiation therapy may shrink the tumor so it can be removed by surgery. Giving docetaxel after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving chemoradiotherapy together with cisplatin and etoposide followed by surgery and docetaxel works in treating patients with newly diagnosed Pancoast tumors, a type of non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of administering induction chemoradiotherapy comprising cisplatin and etoposide followed by surgical resection and adjuvant docetaxel in patients with non-small cell lung cancer involving the superior sulcus (Pancoast tumors).
* Determine overall survival of patients treated with this regimen.
* Determine time to progression in patients treated with this regimen.
* Determine confirmed and unconfirmed and complete and partial response during induction in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE:

* Induction chemoradiotherapy: Patients receive etoposide IV over 1 hour on days 1-5 and 29-33 and cisplatin IV over 1 hour on days 1, 8, 29, and 36. Patients also undergo concurrent radiotherapy once daily 5 days a week for 5 weeks.

Within 2-4 weeks after completion of induction chemoradiotherapy, patients undergo disease evaluation. Patients with no evidence of local or overall disease progression undergo a thoracotomy within 3-7 weeks. Patients who do not qualify for surgery proceed to consolidation chemotherapy within 3-8 weeks after chemoradiotherapy is complete.

* Consolidation chemotherapy: Within 3-8 weeks after thoracotomy, patients with no evidence of disease progression receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4-6 weeks, every 3 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Any of the following stages due to involvement of the superior sulcus:

    * Stage IIB (T3, N0), IIIA (T3, N1), or IIIB (T4, N0-1)
  * Newly diagnosed
  * Primary bronchogenic
* Must meet 1 of the following tumor involvement criteria:

  * An apical tumor associated with the Pancoast syndrome (arm or shoulder pain and/or neurologic findings corresponding to the roots of C-8 and/or T-1 or the inferior trunk of the bronchial plexus with or without Horner's syndrome) without rib or vertebral body involvement
  * Superior sulcus tumors with involvement of the chest wall (T3), usually ribs 1 and 2 by CT scan or MRI, with or without an associated Pancoast syndrome
  * Superior sulcus tumors with invasion of the vertebral bodies or involvement of the subclavian vessels (T4) by CT scan or MRI, with or without an associated Pancoast syndrome
* No more than 1 parenchymal lesion in the same lung or in both lungs
* No involvement of the following lymph node groups as determined by mediastinal exploration* (i.e., mediastinoscopy, mediastinotomy, thoracoscopy, or thoracotomy) within the past 42 days:

  * Single-level or multi-level ipsilateral or contralateral mediastinal nodal (N2 or N3) disease by mediastinoscopy, thoracoscopy, mediastinotomy, thoracotomy, or transbronchial Wang needle biopsy, regardless of whether enlarged nodes are visible or not on chest x-ray or CT scan
  * Supraclavicular (scalene) nodes

    * Any nodes evident on physical exam must be biopsied by fine needle aspiration or open biopsy
  * Left upper lobe tumors with left vocal cord paralysis by indirect laryngoscopy (presumes N2 nodes in the A-P window) NOTE: *Mediastinal exploration is not required for patients whose mediastinum is negative by both positron-emission tomography (PET) and CT scan
* No pleural effusions except if 1 of the following criteria are met:

  * Pleural effusion present before mediastinoscopy or thoracotomy with negative cytology on 2 separate thoracenteses
  * Pleural effusion present only after exploratory or staging thoracotomy, with negative cytology on a single thoracentesis
  * Present only on CT scan and too small to tap
* No pericardial effusions or superior vena cava syndrome
* No brain metastases by CT scan or MRI
* No evidence of distant metastatic disease by bone scan or PET
* Must be a candidate for potential future pulmonary resection

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

  * Patients with Zubrod performance status 2 must have an albumin level at least 0.85 times lower limit of normal and weight loss no greater than 10%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)*
* SGOT or SGPT no greater than 1.5 times ULN* NOTE: *Unless due to a documented benign disease

Renal

* Creatinine clearance at least 50 mL/min

Cardiovascular

* No myocardial infarction within the past 3 months
* No active angina
* No unstable heart rhythms
* No clinically evident congestive heart failure

Pulmonary

* Preresection FEV_1 at least 2.0 L OR
* Predicted postresection FEV_1 greater than 1.0 L

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled peptic ulcer disease
* No grade 2 or greater sensory neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent colony-stimulating factors during chemoradiotherapy or course 1 of consolidation therapy

Chemotherapy

* No prior chemotherapy for lung cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the neck or thorax
* No concurrent intensity-modulated radiotherapy

Surgery

* Prior exploratory thoracotomy allowed only for diagnosis or staging purposes

Other

* No concurrent amifostine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Kraut, MD, Study Chair — Providence Hospital; Tien Hoang, MD, Study Chair — University of Wisconsin, Madison; Valerie W. Rusch, MD, FACS, Study Chair — Memorial Sloan Kettering Cancer Center; James R. Jett, MD, Study Chair — Mayo Clinic; Scott A. Laurie, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre; Alan P. Lyss, MD, Study Chair — Missouri Baptist Cancer Center
Locations (154):
- United States (154):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem: Patients were given induction therapy consisting of concurrent cisplatin + etoposide + 45 Gy thoracic radiation given in 25 daily fractions, followed by thoracotomy, followed by consolidation chemotherapy consisting of three cycles of docetaxel.
Period: Induction Chemotherapy + Radiotherapy
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Started | 46
Completed | 38
Not Completed | 8
Not completed — Ineligible | 1
Not completed — Refused protocol treatment | 1
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 3
Period: Post Chemoradiation Assessment
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Started | 38
Completed | 29
Not Completed | 9
Not completed — Death | 1
Not completed — Disease progression | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Not eligible to continue to surgery | 4
Period: Surgery
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Started | 29
Completed | 22
Not Completed | 7
Not completed — Physician Decision | 4
Not completed — Death | 1
Not completed — Adverse Event | 2
Period: Consolidation Chemotherapy
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Started | 22
Completed | 20
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Number analyzed (Participants) | 44
Age Continuous [Median (Full Range); unit: years] | 59 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Weekly for the first 13 weeks, then every 3 weeks for the next 6 weeks.
Population: Eligible patients who received the study intervention.
Measure: Number; unit: Participants
Arm/Group | Induction Cisplatin/Etoposide + XRT | Surgery | Consolidation Docetaxel
Number analyzed (Participants) | 44 | 29 | 22
Participants
  Adult respiratory distress syndrome (ARDS) | 0 | 3 | 0
  Allergic reaction/hypersensitivity | 1 | 0 | 0
  Chylothorax | 0 | 2 | 0
  Dehydration | 2 | 0 | 2
  Diarrhea | 1 | 0 | 1
  Dyspnea (shortness of breath) | 0 | 0 | 2
  Esophagitis | 1 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 2 | 0 | 1
  Febrile neutropenia | 2 | 0 | 0
  Fistula, pulmonary/upper respiratory - Bronchus | 0 | 1 | 0
  Fistula, pulmonary/upper respiratory - Lung | 0 | 1 | 0
  Glucose, serum-high (hyperglycemia) | 0 | 1 | 1
  Hemoglobin | 3 | 4 | 0
  Hemorrhage/bleeding w/surgery, intra- or post-op | 0 | 1 | 0
  Hypoxia | 0 | 3 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 0 | 1 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Wound | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 0 | 2 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Meninges | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Wound | 0 | 1 | 0
  Infection with unknown ANC - Lung (pneumonia) | 0 | 1 | 0
  Infection with unknown ANC - Wound | 0 | 1 | 0
  Leak, cerebrospinal fluid (CSF) | 0 | 1 | 0
  Leukocytes (total WBC) | 11 | 0 | 6
  Lymphopenia | 3 | 0 | 2
  Metabolic/Laboratory-Other (Specify) | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Esophagus | 1 | 0 | 0
  Nausea | 1 | 0 | 1
  Neutrophils/granulocytes (ANC/AGC) | 15 | 0 | 8
  Pain - Chest wall | 0 | 1 | 0
  Pain - Extremity-limb | 0 | 1 | 0
  Pain-Other (Specify) | 0 | 0 | 1
  Platelets | 0 | 1 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 0 | 1 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 0 | 1 | 0
  Sodium, serum-low (hyponatremia) | 1 | 0 | 0
  Thrombosis/thrombus/embolism | 1 | 0 | 0
  Ventricular arrhythmia - Ventricular fibrillation | 0 | 1 | 0
  Vomiting | 2 | 0 | 1
  Weight loss | 0 | 0 | 1

2. Primary Outcome: Feasibility of Treating Patients With Stage IIB/IIIB Pancoast Tumors With a Regimen of Cisplatin and Etoposide Plus Concurrent Radiotherapy Followed by Surgical Resection Followed by Consolidation Therapy With Docetaxel.
Description: Feasibility was assessed by estimating the percentage of participants who would be able to complete the entire treatment regimen.
Time Frame: After completion of 5 weeks of radiotherapy given concurrently with cisplatin+etoposide, surgery + 8 weeks of recovery time, and 6 weeks of consolidation therapy with docetaxel
Population: Eligible patients who began the treatment regimen were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Number analyzed (Participants) | 44
percentage of participants | 45 [30 to 61]

3. Secondary Outcome: Overall Survival
Description: The duration from the date of enrollment until the date of death due to any cause. Patients last known to be alive were censored at the date of last contact.
Time Frame: daily for 12 weeks then every 3 weeks for 12 weeks, then every 6 months thereafter.
Population: Eligible patients who began the treatment regimen were included in the analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Number analyzed (Participants) | 44
years | 4 [2 to 4]

4. Secondary Outcome: Progression-Free Survival at 3 Years
Description: Duration from date of enrollment to date of progression (per RECIST), symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free were censored at the date of last contact.
Time Frame: At the completion of induction therapy, then again 4 weeks after the completion of consolidation therapy, then every 3 months for 2 years, then every 6 months until up to a maximum of 5 years after enrollment.
Population: Eligible patients who began the treatment regimen were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Number analyzed (Participants) | 44
percentage of patients | 56 [40 to 70]

5. Secondary Outcome: Response
Description: Response was defined as achieving a confirmed or unconfirmed complete or partial response as determined by RECIST. Patients who dropped out due to any cause prior to getting their response assessment were counted as non-responders. A complete response (CR) was defined as disappearance of all disease. A partial response was defined as a >= 30% decrease in the sum of longest diameters of target lesions. A CR or PR was defined as confirmed if two consecutive determinations were documented at least 4 weeks apart.
Time Frame: After completion of induction therapy.
Population: Eligible patients who began the treatment regimen and who had measurable disease (per RECIST) at baseline were included in the analysis of response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Cisplatin/Etoposide + XRT/Surgery/Consolidation Chem
Number analyzed (Participants) | 32
percentage of participants | 28 [14 to 47]

ADVERSE EVENTS:
Time Frame: Weekly for the first 12 weeks, then every 3 weeks for the next 6 weeks.
Arm/Group | Induction Cisplatin/Etoposide + XRT | Surgery | Consolidation Docetaxel
Serious Adverse Events (participants affected / at risk) | 1/44 | 3/29 | 0/22
Other Adverse Events (participants affected / at risk) | 43/44 | 26/29 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Cisplatin/Etoposide + XRT (N=44) | Surgery (N=29) | Consolidation Docetaxel (N=22)
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC - Wound (Infections and infestations) | 0 | 1 | 0
Leukocytes (total WBC) (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Cisplatin/Etoposide + XRT (N=44) | Surgery (N=29) | Consolidation Docetaxel (N=22)
Hemoglobin (Blood and lymphatic system disorders) | 28 | 16 | 13
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0
SVT and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 0 | 2 | 0
SVT and nodal arrhythmia - SVT arrhythmia NOS (Cardiac disorders) | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 17 | 0 | 5
Diarrhea (Gastrointestinal disorders) | 9 | 0 | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 12 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 10 | 0 | 0
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 4 | 0 | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 32 | 0 | 6
Vomiting (Gastrointestinal disorders) | 17 | 0 | 4
Edema: head and neck (General disorders) | 0 | 0 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 32 | 3 | 12
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3 | 5 | 4
Pain-Other (Specify) (General disorders) | 12 | 0 | 7
Rigors/chills (General disorders) | 5 | 0 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Wound (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Wound (Infections and infestations) | 0 | 2 | 0
Rash: dermatitis associated w/radiation (Injury, poisoning and procedural complications) | 16 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 | 0 | 0
AST, SGOT (Investigations) | 4 | 0 | 0
Alkaline phosphatase (Investigations) | 5 | 0 | 2
Creatinine (Investigations) | 0 | 6 | 0
Leukocytes (total WBC) (Investigations) | 24 | 3 | 10
Lymphopenia (Investigations) | 4 | 0 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 19 | 0 | 10
Platelets (Investigations) | 14 | 9 | 0
Weight loss (Investigations) | 11 | 3 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 2 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 0 | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 5 | 4
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 2 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 2 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 | 3 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5
Neuropathy: motor (Nervous system disorders) | 0 | 2 | 0
Neuropathy: sensory (Nervous system disorders) | 9 | 2 | 9
Taste alteration (dysgeusia) (Nervous system disorders) | 12 | 0 | 3
Mood alteration - anxiety (Psychiatric disorders) | 0 | 2 | 0
Mood alteration - depression (Psychiatric disorders) | 3 | 2 | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 | 0 | 3
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No